CLINICAL TRIAL: NCT03010553
Title: Multicenter Phase II Study of Sentinel Node Detection in Squamous Cell Carcinoma T1-T2N0 of the Oropharynx Treated With Radiotherapy and Larynx Treated by Surgery, Laser or Robot
Acronym: GS-OROPHARYNX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-A00922-51; 2006/1217 (Other: CSET number)
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oropharynx (Experimental): Tumors of the oropharynx T1T2N0 treated with radiotherapy
  Interventions: Procedure: Detection and resection of sentinel lymph node
- Larynx (Experimental): Tumors of the T1T2N0 larynx treated by surgery, laser or robot
  Interventions: Procedure: Detection and resection of sentinel lymph node

INTERVENTIONS:
Procedure: Detection and resection of sentinel lymph node

SUMMARY:
Fifty patients with squamous cell carcinoma of the larynx T1 or T2N0 will therefore have a 99mTc lymphoscintigraphy per operative. The identified sentinel node will be removed along with the other lymph nodes of the selective group II and III recess. Sentinel lymph node staging alone and complete dissection with routine anatomical pathology will be compared If this technique is reliable it will make a therapeutic de-escalation in the treatment of small tumors of the larynx by limiting the ganglionic gesture in the patients whose sentinel node is free from metastasis and also to better choose the treatment in case of lymph node involvement

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma T1 or T2 of the oropharynx or larynx, clinical and computed tomography, M0,
2. previously untreated patient, without further concomitant localization,
3. patient over age 18 with no upper age limit, general condition WHO 0 or 1, life expectancy greater than 2 years,
4. on the cervical tomodensitometric assessment with injection of contrast agent: absence of adenomegaly suspicious of metastasis = ganglion of size less than one centimeter and 1.5 cm for group IIa, ovoid, homogeneous, not taking the contrast product And no signs of peri-ganglion invasion (fatty hyperdensity, vascular adhesion), absence of ganglionic grouping (> 3)
5. Untreated patient outside a biopsy excision (melanoma experiment),
6. Possibility of realizing an IMRT
7. Informing the patient and signing informed consent.

Exclusion Criteria:

1) Patient already treated for this tumor outside a biopsy excision, 2) Contraindications to radiotherapy, scintigraphy or procedure, allergy to Rhenium sulphide or 99m Technetium 3) History of epidermoid carcinoma of VADS 4) Pregnant woman, likely to be pregnant or nursing, (5) Persons deprived of their liberty or under guardianship, 6) Impossibility to submit to the medical follow-up of the trial for geographical, social or psychological reasons.

7) Patient who underwent cervical surgery for any cause 8) Patient with cervical radiotherapy 9) Patient unable to undergo cervical lymph node dissection 10) Patient treated for another cancer outside the VADS within a period of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reliability of the sentinel lymph node technique | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No